CLINICAL TRIAL: NCT05684185
Title: Immunogenicity Assessment of Subjects Receiving Rabies Post-exposure Prophylaxis in Cambodia
Status: Completed | Type: Observational
Sponsor: Institut Pasteur du Cambodge (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: RAB00056
Record Dates: First submitted 2022-10-16; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Rabies Post-exposure Prophylaxis
MeSH Terms: interventions — Injections, Intramuscular; Injections, Intradermal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- IM, <15 years old: Group with Intramuscular (IM) rabies post-exposure prophylaxis
  Interventions: Biological: Intramuscular (IM) rabies post-exposure prophylaxis
- IM, 15 years old and older: Group with Intramuscular (IM) rabies post-exposure prophylaxis
  Interventions: Biological: Intramuscular (IM) rabies post-exposure prophylaxis
- ID, <15 years old: Group with Intradermal (ID) rabies post-exposure prophylaxis
  Interventions: Biological: Intradermal (ID) rabies post-exposure prophylaxis
- ID, 15 years old and older: Group with Intradermal (ID) rabies post-exposure prophylaxis
  Interventions: Biological: Intradermal (ID) rabies post-exposure prophylaxis

INTERVENTIONS:
Biological: Intramuscular (IM) rabies post-exposure prophylaxis — one-site, 0.5 mL at Day 0, D3, D7 and D14
  Groups: IM, 15 years old and older; IM, <15 years old
Biological: Intradermal (ID) rabies post-exposure prophylaxis — two-site, 0.1 mL at Day 0, D3 and D7
  Groups: ID, 15 years old and older; ID, <15 years old

SUMMARY:
A rabies virus neutralizing antibody (RVNA) concentration ≥ 0.5 IU/ml at 14 days after immunization is considered a proxy for protection in vaccine efficacy studies. Abridged and dose-sparing vaccination regimens increase accessibility and reduce both direct and indirect costs, especially in resource-constrained countries where RABV prevalence is highest. Several efficacy studies evaluated safety and immunogenicity of abridged regimens in healthy adult volunteers using either four-site intradermal (ID) or intramuscular (IM) regimens, showing them to be safe and immunogenic.

Researchers at the Institut Pasteur du Cambodge (IPC) have previously conducted a retrospective study on clinical outcome at ≥6 months in 3318 Cambodians who received intradermal Vero cell vaccine post-exposure prophylaxis after a bite by a rabid or sick-looking but untested dog in 2003-2014. Here, the investigators could show that there was no significant difference in survival among patients who received 3 versus 4 sessions of the Thai Red Cross (TRC) ID regimen. In a separate study, investigators measured antibody responses in order to evaluate the immunogenicity of the TRC regiment after 3 sessions versus 4 sessions. The investigators did not observe an increase in rabies virus seroneutralization titers 14 days after the fourth immunization compared to 14 days after the third immunization. These results contributed to changes endorsed by the WHO in its April 2018 guidelines. The "Institut Pasteur du Cambodge (IPC) regimen" of three PEP sessions of two-site ID 0.1 mL vaccine doses each at days 0, 3 and 7 is the first one-week PEP regimen to be recommended.

In the current research project, the aim is to compare further different PEP vaccination strategies in a real life setting of individuals attending the rabies vaccination center at Institut Pasteur du Cambodge (IPC) in Phom Penh, Cambodia. The antibody kinetics and cellular immune responses in patients following either the one-week, 2-site ID regimen (IPC regimen) or the two-week IM regimen (4-dose regimen) as well as the participants' survival for both protocols after 6 months are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects entering a rabies post-exposure vaccination course whatever the vaccine used with or without administration of rabies immunoglobulin (RIGs).
* Subjects with ability to attend all scheduled visits and to comply with all study procedures

Exclusion Criteria:

* Subjects with history of previous rabies vaccination

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients seeking for rabies post-exposure prophylaxis (PEP) at the rabies prevention center of Institut Pasteur du Cambodge
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Changes of the level of rabies virus neutralizing antibodies at 14 days and 18 days after first dose among patients receiving post-exposure prophylaxis (PEP) using intramuscular (IM) and intradermal (ID) protocols | Day 0 (the first PEP dose), then 14 days and 28 days after Day 0 in each study group (IM / ID)
  Assessment of humoral immune response (rabies virus neutralizing antibodies - RVNA - titers measured with Fluorescent Antibody Virus Neutralization test - FAVN - by local laboratory) at different time points: at baseline before the first PEP dose, 14 days and 28 days after the first PEP dose, in each study group (IM / ID)

CONTACTS AND LOCATIONS:
Overall Officials: Sowath LY, PhD, Principal Investigator — Institut Pasteur du Cambodge (IPC)
Locations (1):
- Institut Pasteur du Cambodge (IPC), Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: Undecided